CLINICAL TRIAL: NCT05290766
Title: Two Versus Four Implant Supporting Fixed Full-arch Screw-retained Metal Acrylic Hybrid Mandibular Prosthesis.(A Study of Patient Satisfaction)
Brief Title: Two Versus Four Implant-supported Fixed Full-arch Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A03040122
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2023-04

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): will receive implant-supported mandibular fixed metal acrylic prosthesis on 4 implants that were placed according to the "All on four concept".
  Interventions: Procedure: placement of four dental implants; Device: mandibular full arch prosthesis
- Study group (Active Comparator): will receive implant-supported mandibular fixed metal acrylic prosthesis on two implants placed according to "All On two concept".
  Interventions: Procedure: placement of two dental implants; Device: mandibular full arch prosthesis

INTERVENTIONS:
Procedure: placement of four dental implants — placement of four dental implants according to the " All on four concept"
  Arms: Control group
Procedure: placement of two dental implants — placement of two dental implants according to " All on two concepts"
  Arms: Study group
Device: mandibular full arch prosthesis — loading of the mandibular fixed full-arch screw-retained metal acrylic prosthesis

SUMMARY:
The aim of this study will be the evaluation of patient satisfaction and oral health-related-quality of life (OHRQoL) of two versus four implants supporting fixed full-arch screw-retained metal acrylic hybrid mandibular prosthesis.

DETAILED DESCRIPTION:
* Six completely edentulous patients will be selected for this study from the outpatient clinic of the prosthodontic department
* All patients will be informed about all surgical and prosthodontics procedures that will be done for them. All patients will sign the consent form of the ethical committee in faculty dentistry Mansoura University.

The patients will be divided into 2 groups

1. Control group: will receive implant-supported mandibular fixed metal acrylic prosthesis on 4 implants that were placed according to the "All on four concept".
2. Study group: will receive implant-supported mandibular fixed metal acrylic prosthesis on two implants placed according to "All On two concept".

ELIGIBILITY:
Inclusion Criteria:

* • Eligible patients needed must have Sufficient interarch space (at least 15 mm from the occlusal plane to the mandibular ridge) to provide space for fixed prosthesis construction all patients should be completely edentulous patients with resorbed mandibular ridge all patients must be angle class I

Exclusion Criteria:

* systemic diseases that contraindicate implant placement bone metabolic diseases such as diabetes mellitus irradiation of the head and neck region chemotherapy within the past 3 years smoking habits.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2023-04-16 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) questionnaire | one year
  Regarding VAS, participants were asked to score their answer according to the amount of satisfaction on a 100mm line (Score zero = no satisfaction at all and score 100 = complete satisfaction). The questions cover several items related to prosthesis such as: retention, stability, comfort, ease of cleaning, ease of speaking, ease of chewing, limited activities due to embarrassment, quality of bolus and appearance

SECONDARY OUTCOMES:
Quality of Life (Secondary Outcome). | one year
  The oral Health impact profile (OHIP-14) questions were utilized to assess OHRQoL. The questions were composed of seven domains

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Dentistry, Mansoura University, Al Mansurah, Eldakahlia
  - Christine Ibrahim, Al Mansurah

IPD SHARING:
Plan to Share IPD: No